CLINICAL TRIAL: NCT01886755
Title: Efficacy of an Oral Rehydration Solution Containing the Probiotic Lactobacillus Reuteri Protectis and Zinc in Infants With Acute Gastroenteritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandra Papadopoulou (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Sponsor-Investigator, Alexandra Papadopoulou, Consultant Pediatrician, Aghia Sophia Children's Hospital of Athens
Organization: Aghia Sophia Children's Hospital of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CSUB0069
Record Dates: First submitted 2013-06-22; First posted 2013-06-26 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Acute Gastroenteritis
Keywords: Acute gastroenteritis; Probiotics; Lactobacillus reuteri; Zinc supplementation; Infants; Age 6 months to 36 months
MeSH Terms: interventions — World Health Organization oral rehydration solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ORS with probiotic and zinc (Experimental): ORS with probiotic and zinc Oral rehydration solution with freeze-dried Lactobacillus reuteri DSM 17938 and zinc sulphate
  Interventions: Dietary Supplement: ORS rehydration solution
- Placebo Comparator (Placebo Comparator): Standard oral rehydration solution
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: ORS rehydration solution
  Arms: ORS with probiotic and zinc
Dietary Supplement: placebo
  Arms: Placebo Comparator

SUMMARY:
An ORS with L. reuteri DSM 17938 and zinc is expected to reduce duration and severity of symptoms in infants and young children with acute gastroenteritis.

DETAILED DESCRIPTION:
Oral rehydration solution is recommended for treatment and prevention of dehydration due to acute gastroenteritis in infants and children (WHO/UNICEF, 2004; ESPGHAN / ESPID Guidelines, 2008). Acute diarrhoea may lead to zinc depletion in infants, and zinc supplementation is recommended in infants and children with acute gastroenteritis living in developing countries. In developed countries however, the studies on the efficacy of zinc supplementation in children with acute gastroenteritis are few and conflicting.

Selected strains of probiotics, including L. reuteri ATCC 55730, have been shown in several studies to reduce the duration and the severity of diarrhoea in children with acute gastroenteritis and the effect is greater if the probiotics are given within 60 hours from the onset of symptoms. Lactobacillus reuteri (L. reuteri) has been shown to reduce the duration and severity of acute gastroenteritis in children aged 6-36 months. In these studies L. reuteri was reported to have clinical effect on diarrhoea of both bacterial and viral (rotavirus) origin. Furthermore, L. reuteri strain DSM 17938 has recently been shown to reduce the duration of watery diarrhoea by 1.2 days among 6-36 mo old Italian children with acute gastroenteritis treated in hospital.

The present study is a prospective, randomized, double blind, controlled study with parallel groups. The planned investigation is designed to compare the efficacy of an ORS with L. reuteri DSM 17938 and zinc to an ORS with similar osmolarity and content of salts but without L. reuteri DSM 17938 and zinc, on the duration and severity of acute gastroenteritis. 92 children aged 6-36 months seen at private pediatric clinics and/or at the emergency clinics of the Athens Childrens Hospital "AGIA SOPHIA", and treated either as outpatients or as inpatients will be recruited until the final sample size is reached. Assuming a difference of 30% between groups in the primary outcome of prevalence of diarrhoea on day 2, and estimating an attrition rate of approximately 15%, the final sample size will be 92 subjects, or 46 subjects in each arm.

Data collection points will be on day 7 at the outpatient clinic of the Division of Pediatric Gastroenterology & Nutrition of the First Department of Paediatrics, Athens University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* 6 - 36 months old children
* 3 or more watery or soft stools per day for the past 24-48 hours
* Clinically judged as having mild to moderate dehydration (Bailey scale scores 1 to 4)
* Available throughout the study period
* Re-examination on the 7th day from the enrolment
* The signed informed consent by one/both parents or legal guardian
* Parents or legal guardian should have the mental ability to understand and willingness to fulfil all the details of the protocol

Exclusion Criteria:

* Diarrhoea lasting more than 48 h
* Clinical signs of severe dehydration (Bailey scale scores = or > 5)
* Malnutrition as judged by a body weight/height ratio below the 5th percentile
* Clinical signs of a coexisting severe acute systemic illness (meningitis, sepsis, pneumonia)
* Immunodeficiency
* Severe chronic disease including cystic fibrosis
* Food allergy diagnosed by physician or other chronic gastrointestinal diseases
* Use of pre-/probiotics in the previous 2 weeks, for example infant formula containing probiotics and/or prebiotics.
* Use of antibiotics or any anti-diarrhoeal medication in the previous 4 weeks

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 51 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Resolution of diarrhoea. | 48 hrs after start of treatment
  1. Proportion of children without watery (3A ISS by Amsterdam infant stool scale ) or soft (3B ISS Amsterdam infant stool scale) stools on day 2 of treatment. Day 0 = day of enrolment and start of treatment, day 1 = first complete day of treatment
  2. Time from start of treatment and until last watery or soft stool.

SECONDARY OUTCOMES:
Reduction of severity of diarrhoea | 120 hrs from the start on treatment
  Reduction of severity of diarrhoea will be evaluated as though :
  1. Number of watery (type 3A ISS ) and soft ( 3B ISS) stools daily on each of the day of the therapy and up to 5 days.
  2. Proportion of children with watery (3A ISS) and soft ( 3B ISS) stools on each of the day 1-5 (Day 0 = day of enrolment and start of treatment, day 1 = first complete day of treatment)
     * Νumber of vomiting episodes: per child on each of the treatment days 1-5.
     * Volume of ORS intake during the first 24h of treatment.
     * Need of hospitalization
     * Absence of workdays for the parents.
     * Child's absence from day care / nursery.
     * Medication needed for treatment of diarrhoea.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Papadopoulou, Dr, Principal Investigator — Athens Children's Hospital "AGIA SOPHIA"
Locations (1):
- Athens Children's Hospital "AGIA SOPHIA", Athens, Attica, Greece